CLINICAL TRIAL: NCT00272688
Title: Continuous Delivery of Levodopa/Carbidopa (Duodopa) in Patients With Advanced Idiopathic Parkinsons Disease - a Health Economic Evaluation
Brief Title: Continuous Delivery of Levodopa in Patients With Advanced Idiopathic Parkinsons Disease - Cost-benefit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Christofer Lundqvist, Principal investigator, University Hospital, Akershus
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Duo-HRQoL-2
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Levodopa (drug), intraduodenal administration

SUMMARY:
An open, observational health economic study to estimate marginal cost and health consequences of replacing conventional Parkinsons disease therapy with intraduodenal levodopa administered continuously

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of of idiopathic Parkinsons disease
* Motor fluctuations despite optimised per oral treatment

Exclusion Criteria:

* Severe dementia, confusion, psychosis or depression
* Patients with contraindications against levodopa treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Marginal cost per QALY of replacing conventional treatment with intraduodenal levodopa | one year
Quality of life at three, six, nine and twelve months(Assessed by Nottingham Health Profile (NHP), Parkinson Disease Questionnaire (PDQ39), 15D Quality of life)

SECONDARY OUTCOMES:
Parkinson related function at three, six, nine and twelve months(UPDRS, Hoehn and Yahr scores, Schwab and England)

CONTACTS AND LOCATIONS:
Overall Officials: Christofer Lundqvist, PhD, M.D., Principal Investigator — HØKH - Helse Ost Health Services Research Centre, Akershus University Hospital, Norway; Antonie Beiske, PhD, M.D., Principal Investigator — Dept Neurology, Akershus University Hospital, Norway
Locations (2):
- Norway (2):
  - Akershus University Hospital, Nordbyhagen
  - Dept Neurology, Ulleval University Hospital, Oslo